CLINICAL TRIAL: NCT00150800
Title: An Open-label, Multi-center, Follow-up Trial to Evaluate Long Term Safety and Efficacy of Brivaracetam Used as Adjunctive Treatment at a Flexible Dose up to a Maximum of 200 mg/Day in Subjects Aged 16 Years or Older Suffering From Epilepsy
Brief Title: This Trial, Evaluating the Long-term Safety and Tolerability of Brivaracetam Will Provide Subjects Suffering From Epilepsy, Who May Have Benefited From Brivaracetam as Adjunctive Treatment, the Opportunity to Receive Open Label Brivaracetam Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB PHARMA Inc. (US) (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01199
Expanded Access: NCT03532516 (Available)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Epilepsy
Keywords: Brivaracetam; Epilepsy; Partial Onset Seizures; open label
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brivaracetam (Experimental): Brivaracetam used as adjunctive treatment, flexible dosing up to 200 mg /day in b.i.d (twice daily) administration. Dose increase or decrease can be made in increments of maximum 50 mg/day on a weekly basis.
  Interventions: Drug: Brivaracetam

INTERVENTIONS:
Drug: Brivaracetam — * Active Substance: Brivaracetam
  * Pharmaceutical Form: Tablet
  * Concentration: 10 mg and 25 mg
  * Route of Administration: Oral

SUMMARY:
This trial, evaluating the long-term safety and tolerability of brivaracetam will provide subjects suffering from epilepsy, who may have benefited from brivaracetam as adjunctive treatment, the opportunity to receive open label brivaracetam treatment.

DETAILED DESCRIPTION:
Study access was limited to subjects having completed one of the previous brivaracetam (BRV) studies: N01193 [NCT00175825], N01252 [NCT00490035], N01253 [NCT00464269], N01254 [NCT00504881].

ELIGIBILITY:
Inclusion Criteria:

* Male/ female subjects from 16 years and on. Subjects under 18 years may only be included where legally permitted and ethically accepted
* Subjects with epilepsy who have participated in previous brivaracetam trials which allow access to the present study
* Subjects for whom the investigator believes a reasonable benefit from the long term administration of brivaracetam may be expected
* Female subjects without childbearing potential. Female subjects with child bearing potential are eligible if they use a medically accepted contraceptive method for the duration of the study
* Subject/ legally acceptable representative considered as reliable and capable of adhering to the protocol, visit schedule or medication intake according to the judgment of the Investigator

Exclusion Criteria:

* Severe medical, neurological and psychiatric disorders or laboratory values which may have an impact on the safety of the subject
* Poor compliance with the visit schedule or medication intake in the previous brivaracetam study
* Pregnant or lactating women
* Participation in any clinical study of another investigational drug or device during the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2006-01; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (100):
- United States (46):
  - N01199 1051, Phoenix, Arizona
  - N01199 1362, Phoenix, Arizona
  - N01199 1374, Tucson, Arizona
  - N01199 1050, Little Rock, Arkansas
  - N01199 1078, Fresno, California
  - N01199 1392, Newport Beach, California
  - N01199 1087, San Francisco, California
  - N01199 1368, San Francisco, California
  - N01199 1396, Atlanta, Georgia
  - N01199 1385, Augusta, Georgia
  - N01199 1356, Chicago, Illinois
  - N01199 1388, Springfield, Illinois
  - N01199 1375, Wichita, Kansas
  - N01199 1364, Lexington, Kentucky
  - N01199 1380, Louisville, Kentucky
  - N01199 1052, Paducah, Kentucky
  - N01199 1083, Ruston, Louisiana
  - N01199 1373, Baltimore, Maryland
  - N01199 1086, Bethesda, Maryland
  - N01199 1077, Burlington, Massachusetts
  - N01199 1391, Detroit, Michigan
  - N01199 1395, Detroit, Michigan
  - N01199 1071, Grand Rapids, Michigan
  - N01199 1389, Saint Paul, Minnesota
  - N01199 1079, Tupelo, Mississippi
  - N01199 1360, Chesterfield, Missouri
  - N01199 1352, St Louis, Missouri
  - N01199 1069, Great Falls, Montana
  - N01199 1062, Toms River, New Jersey
  - N01199 1053, New York, New York
  - N01199 1365, Rochester, New York
  - N01199 1366, Cincinnati, Ohio
  - N01199 1054, Columbus, Ohio
  - N01199 1359, Portland, Oregon
  - N01199 1055, Philadelphia, Pennsylvania
  - N01199 1059, Philadelphia, Pennsylvania
  - N01199 1081, Greenville, South Carolina
  - N01199 1061, Nashville, Tennessee
  - N01199 1084, Dallas, Texas
  - N01199 1394, Dallas, Texas
  - N01199 1064, Houston, Texas
  - N01199 1082, Salt Lake City, Utah
  - N01199 1367, Charlottesville, Virginia
  - N01199 1393, Richmond, Virginia
  - N01199 1376, Seattle, Washington
  - N01199 1369, Milwaukee, Wisconsin
- Australia (8):
  - N01199 1420, Chatswood, New South Wales
  - N01199 1430, Randwick, New South Wales
  - N01199 1423, Adelaide, South Australia
  - N01199 1428, Woodville, South Australia
  - N01199 1427, Clayton, Victoria
  - N01199 1426, Parkville, Victoria
  - N01199 1421, West Heidelberg, Victoria
  - N01199 1422, Fitzroy
- Brazil (13):
  - N01199 1028, Campinas
  - N01199 1325, Curitiba
  - N01199 1024, Florianópolis
  - N01199 1150, Florianópolis
  - N01199 1331, Porto Alegre
  - N01199 1332, Porto Alegre
  - N01199 1022, Riberao Preto
  - N01199 1023, Salvador
  - N01199 1029, São José do Rio Preto
  - N01199 1021, São Paulo
  - N01199 1027, São Paulo
  - N01199 1030, São Paulo
  - N01199 1326, São Paulo
- Canada (5):
  - N01199 1316, Edmonton, Alberta
  - N01199 1312, Greenfield Park, Quebec
  - N01199 1311, Montreal, Quebec
  - N01199 1314, Montreal, Quebec
  - N01199 1313, Québec, Quebec
- India (18):
  - N01199 1266, Mumbai, Maharashti
  - N01199 1045, Bangalore
  - N01199 1256, Bangalore
  - N01199 1257, Bangalore
  - N01199 1261, Bangalore
  - N01199 1046, Chennai
  - N01199 1042, Hyderabad
  - N01199 1253, Hyderabad
  - N01199 1262, Hyderabad
  - N01199 1258, Jaipur
  - N01199 1040, Lucknow
  - N01199 1250, Lucknow
  - N01199 1043, Mumbai
  - N01199 1259, Mumbai
  - N01199 1265, Parel Mumbai
  - N01199 1251, Pune
  - N01199 1264, Pune Maharashtra
  - N01199 1263, Tirupati
- Mexico (10):
  - N01199 1412, San Nicholas de Los Garza, Nuevo León
  - N01199 1010, Aguascalientes
  - N01199 1008, Chihuahua City
  - N01199 1009, Chihuahua City
  - N01199 1003, Guadalajara
  - N01199 1403, Mexico City
  - N01199 1005, Monterrey
  - N01199 1007, Monterrey
  - N01199 1002, San Luis Potosí City
  - N01199 1001, Zapopan

REFERENCES:
- [Result] O'Brien TJ, Borghs S, He QJ, Schulz AL, Yates S, Biton V. Long-term safety, efficacy, and quality of life outcomes with adjunctive brivaracetam treatment at individualized doses in patients with epilepsy: An up to 11-year, open-label, follow-up trial. Epilepsia. 2020 Apr;61(4):636-646. doi: 10.1111/epi.16484. Epub 2020 Mar 28. PMID 32221987
- [Result] Moseley BD, Dimova S, Elmoufti S, Laloyaux C, Asadi-Pooya AA. Long-term efficacy and tolerability of adjunctive brivaracetam in adults with focal to bilateral tonic-clonic (secondary generalized) seizures: Post hoc pooled analysis. Epilepsy Res. 2021 Oct;176:106694. doi: 10.1016/j.eplepsyres.2021.106694. Epub 2021 Jun 24. PMID 34218211
- [Derived] Markham A. Brivaracetam: First Global Approval. Drugs. 2016 Mar;76(4):517-22. doi: 10.1007/s40265-016-0555-6. PMID 26899665

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in January 2006 and concluded in September 2017. 668 subjects were included in the Enrolled Set but 1 subject from India lost to follow up and was excluded from the Safety Analysis Set due to lack of medical data.
Pre-assignment Details: The Participant Flow refers to the Safety Analysis Set which included all subjects who took at least 1 dose of study drug.
Groups:
- Brivaracetam: Brivaracetam (BRV) used as adjunctive treatment, flexible dosing up to 200 mg /day in b.i.d (twice daily) administration. Dose increase or decrease can be made in increments of maximum 50 mg /day on a weekly basis.
Period: Overall Study
Arm/Group | Brivaracetam
Started | 667
Completed | 171
Not Completed | 496
Not completed — Adverse Event | 89
Not completed — Death | 18
Not completed — Lack of Efficacy | 166
Not completed — Lost to Follow-up | 58
Not completed — Subject's choice | 90
Not completed — No compliance | 18
Not completed — IP misshandling | 1
Not completed — Site closure | 24
Not completed — Protocol non-adherence | 2
Not completed — Nobody to accompany patient | 1
Not completed — Distance too long for patient | 1
Not completed — Neurosurgery | 2
Not completed — BRV monotherapy | 1
Not completed — Visit refusal | 3
Not completed — Sponsor's request | 2
Not completed — Generalized Epilepsy | 1
Not completed — Moved from area/country | 8
Not completed — PI retiring | 2
Not completed — PI leaving site | 2
Not completed — Patient insurance | 1
Not completed — Surgical intervention | 4
Not completed — Pregnancy planned | 1
Not completed — PI discontinuation request | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Characteristics refers to the Safety Analysis Set which included all subjects who took at least 1 dose of study drug.
Arm/Group | Brivaracetam
Number analyzed (Participants) | 667
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 632
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 303
  Male | 364
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 21
  Asian | 206
  Black | 18
  Native Hawaiian Or Other Pacific Islander | 1
  White | 361
  Other/Mixed | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Treatment-Emergent Adverse Event (TEAE) During the Study Period
Description: Treatment-Emergent Adverse Events (TEAEs) are any untoward medical incidence in a subject during administered study treatment, whether or not these events are related to study treatment.
Time Frame: Visit 1 through last Evaluation Period, Down-Titration, or Post-Treatment Periods (up to 11 years)
Population: The Safety Analysis Set consisted of all subjects who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Brivaracetam (SS): Brivaracetam (BRV) used as adjunctive treatment, flexible dosing up to 200 mg /day in b.i.d (twice daily) administration. Dose increase or decrease can be made in increments of maximum 50 mg /day on a weekly basis.
Arm/Group | Brivaracetam (SS)
Number analyzed (Participants) | 667
percentage of participants | 91.2

2. Primary Outcome: Percentage of Participants Who Withdrew Due to an Adverse Event (AE) During the Study Period
Description: Adverse Events (AE) are any untoward medical incidence in a subject during administered study treatment, whether or not these events are related to study treatment.
Time Frame: Visit 1 through last Evaluation Period, Down-Titration, or Post-Treatment Periods (up to 11 years)
Population: The Safety Analysis Set consisted of all subjects who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Brivaracetam (SS)
Number analyzed (Participants) | 667
percentage of participants | 14.8

3. Primary Outcome: Percentage of Participants With a Serious Adverse Event (SAE) During the Study Period
Description: A Serious Adverse Event (SAE) is any untoward medical incidence that occurs at any dose.
Time Frame: Visit 1 through last Evaluation Period, Down-Titration, or Post-Treatment Periods (up to 11 years)
Population: The Safety Analysis Set consisted of all subjects who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Brivaracetam (SS)
Number analyzed (Participants) | 667
percentage of participants | 22.8

4. Secondary Outcome: Partial Onset Seizure (POS) (Type I) Frequency Per 28 Days During the Evaluation Period
Description: Baseline is the Baseline from subject's previous study of enrollment period. N01193 [NCT00175825], N01252 [NCT00490035], N01253 [NCT00464269], N01254 [NCT00504881].
  A 28 day Type 1 seizure frequency is the total number of Type 1 seizures divided by the total number of days evaluated multiplied by 28.
Time Frame: From Baseline of the previous study to the Evaluation Period (up to 11 years)
Population: The Partial Onset Seizure (POS) Efficacy Analysis Set consisted of all subjects with POS who took at least 1 dose of study drug and had at least 1 seizure diary day during the Evaluation Period.
Measure: Median (Inter-Quartile Range); unit: Seizures per 28 days
Groups:
- Brivaracetam (POS-ES): Brivaracetam (BRV) used as adjunctive treatment, flexible dosing up to 200 mg /day in b.i.d (twice daily) administration. Dose increase or decrease can be made in increments of maximum 50 mg /day on a weekly basis.
Arm/Group | Brivaracetam (POS-ES)
Number analyzed (Participants) | 648
Seizures per 28 days
  baseline | 9.2 [5.5 to 20.2]
  on treatment | 4.2 [1.6 to 11.3]

5. Secondary Outcome: Percent Change in Partial Onset Seizure (POS) (Type I) Frequency Per 28 Days From Baseline of the Previous Study to the Evaluation Period
Description: The percent change from the previous study baselines, in Partial Onset Seizure (POS) (Type I) frequency per 28 days is defined as:
  (the value at the previous study baselines) minus (the value at each time-points during the evaluation period) divided by the value at the previous study baselines.
Time Frame: From Baseline of the previous study to the Evaluation Period (up to 11 years)
Population: The Partial Onset Seizures (POS) Efficacy Analysis Set consisted of all subjects with POS who took at least 1 dose of study drug and had at least 1 seizure diary day during the Evaluation Period.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Brivaracetam (POS-ES)
Number analyzed (Participants) | 648
percent change | 57.3 [18.6 to 82.2]

6. Secondary Outcome: Percentage of Participants With Response for Partial Onset Seizure (POS) (Type I) Frequency Over the Evaluation Period
Description: A responder is defined as a subject with a higher than or equal to (>=) 50 % change in seizure frequency from Baseline period of the previous study.
Time Frame: From Baseline of the previous study to the Evaluation Period (up to 11 years)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Brivaracetam (POS-ES)
Number analyzed (Participants) | 648
percentage of participants | 55.6

ADVERSE EVENTS:
Time Frame: Visit 1 through last Evaluation Period, Down-Titration, or Post-Treatment Periods (up to 11 years)
Arm/Group | Brivaracetam
All-Cause Mortality (participants affected / at risk) | 18/667
Serious Adverse Events (participants affected / at risk) | 152/667
Other Adverse Events (participants affected / at risk) | 521/667
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam (N=667)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 1 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastric fistula (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Splenic artery aneurysm (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 2 (3)
Drug ineffective (General disorders) | 1 (2)
Multi-organ failure (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (2)
Pyrexia (General disorders) | 2 (2)
Sudden unexplained death in epilepsy (General disorders) | 2 (2)
Unevaluable event (General disorders) | 3 (3)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (3)
Cellulitis staphylococcal (Infections and infestations) | 1 (1)
Coccidioidomycosis (Infections and infestations) | 1 (1)
Dengue fever (Infections and infestations) | 2 (2)
Disseminated tuberculosis (Infections and infestations) | 1 (1)
Encephalitis herpes (Infections and infestations) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Malaria (Infections and infestations) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1)
Meningitis tuberculous (Infections and infestations) | 1 (3)
Neurocysticercosis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 7 (9)
Pyelonephritis (Infections and infestations) | 1 (1)
Rickettsiosis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Viral infection (Infections and infestations) | 1 (1)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (3)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 4 (4)
Ulna fracture (Injury, poisoning and procedural complications) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Anticonvulsant drug level increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ocular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Ataxia (Nervous system disorders) | 2 (2)
Central nervous system lesion (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 3 (3)
Complicated migraine (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 15 (20)
Dizziness (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Partial seizures (Nervous system disorders) | 2 (2)
Postictal state (Nervous system disorders) | 2 (2)
Seizure cluster (Nervous system disorders) | 1 (2)
Somnolence (Nervous system disorders) | 2 (2)
Status epilepticus (Nervous system disorders) | 6 (7)
Transient ischaemic attack (Nervous system disorders) | 4 (4)
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 5 (5)
Pregnancy on contraceptive (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Pregnancy on oral contraceptive (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 1 (1)
Aggression (Psychiatric disorders) | 2 (2)
Completed suicide (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Schizophrenia (Psychiatric disorders) | 1 (1)
Self-injurious ideation (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 2 (2)
Suicide attempt (Psychiatric disorders) | 7 (8)
Calculus ureteric (Renal and urinary disorders) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 2 (2)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Scrotal disorder (Reproductive system and breast disorders) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Abortion induced (Surgical and medical procedures) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam (N=667)
Nausea (Gastrointestinal disorders) | 67 (93)
Diarrhoea (Gastrointestinal disorders) | 65 (86)
Vomiting (Gastrointestinal disorders) | 58 (109)
Toothache (Gastrointestinal disorders) | 42 (66)
Abdominal pain (Gastrointestinal disorders) | 39 (55)
Constipation (Gastrointestinal disorders) | 38 (48)
Pyrexia (General disorders) | 69 (132)
Fatigue (General disorders) | 51 (63)
Irritability (General disorders) | 42 (50)
Nasopharyngitis (Infections and infestations) | 94 (154)
Influenza (Infections and infestations) | 84 (177)
Upper respiratory tract infection (Infections and infestations) | 76 (137)
Urinary tract infection (Infections and infestations) | 64 (150)
Fall (Injury, poisoning and procedural complications) | 40 (72)
Contusion (Injury, poisoning and procedural complications) | 34 (68)
Laceration (Injury, poisoning and procedural complications) | 34 (65)
Decreased appetite (Metabolism and nutrition disorders) | 36 (41)
Back pain (Musculoskeletal and connective tissue disorders) | 64 (88)
Arthralgia (Musculoskeletal and connective tissue disorders) | 52 (66)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 44 (63)
Headache (Nervous system disorders) | 165 (420)
Dizziness (Nervous system disorders) | 142 (254)
Somnolence (Nervous system disorders) | 91 (116)
Convulsion (Nervous system disorders) | 70 (99)
Tremor (Nervous system disorders) | 38 (48)
Depression (Psychiatric disorders) | 70 (85)
Insomnia (Psychiatric disorders) | 49 (65)
Anxiety (Psychiatric disorders) | 45 (65)
Cough (Respiratory, thoracic and mediastinal disorders) | 46 (69)
Rash (Skin and subcutaneous tissue disorders) | 34 (56)
Hypertension (Vascular disorders) | 46 (55)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-10-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT00150800/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT00150800/SAP_001.pdf